CLINICAL TRIAL: NCT00078507
Title: Sensory Re-Training Following Orthognathic Surgery
Brief Title: Sensory Re-Training Following Facial Surgery for Correction of Facial Skeletal Disharmony
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDCR-13967; R01DE013967 (NIH)
Record Dates: First submitted 2004-03-01; First posted 2004-03-03 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Mandibular Advancement
Keywords: Outcome and Process Assessment (Health Care); Behavior Control; Sensation; Randomized Controlled Trials; Adolescent; Adult

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Opening Exercises Only (Active Comparator): Standard of care opening exercises following BSSO surgery to regain mouth opening
  Interventions: Behavioral: Opening Exercises
- Sensory Retraining Exercises (Experimental): 3 sets of facial exercises performed with soft cosmetic brush 1 wk - 4 wks after surgery; 4wks to 3 mos after surgery; 3 mos to 6 mos after surgery.
  Interventions: Behavioral: Sensory Re-training; Behavioral: Sensory Retraining

INTERVENTIONS:
Behavioral: Sensory Re-training
  Arms: Sensory Retraining Exercises
Behavioral: Sensory Retraining — Facial Exercises
  Arms: Sensory Retraining Exercises
Behavioral: Opening Exercises
  Arms: Opening Exercises Only

SUMMARY:
The purpose of this study is to determine whether facial exercises in conjunction with opening exercises routinely provided after facial surgery to correct a facial skeletal disharmony will shorten the time until a patient receives no unpleasant or negative facial sensation.

DETAILED DESCRIPTION:
Abnormal facial sensation has a negative impact on patients' oral behaviors and may adversely affect a patient's quality of life if the altered sensation persists. Many patients with abnormal sensations retain some sensory function and do not develop chronic pain, and for those individuals there are currently no evidence-based noninvasive therapies. The goal of this project is to evaluate sensory re-training, a rehabilitative therapy that offers significant potential for patients who experience impaired sensory function regardless of the cause. This behavioral therapy approach has been used with substantial clinical success with hand injury patients since the 1970s. Re-training appears to enhance central reorganization of impulses from an injured sensory nerve to the cerebral cortex so that the altered sensory signals can be interpreted and translated into functionally meaningful motor functions.

Sensory re-training will be compared to a placebo jaw-opening exercise in a single blind, randomized two-arm parallel group stratified block clinical trial, using orthognathic surgery patients as subjects. Orthognathic surgery patients offer an uncompromised model for the evaluation of new rehabilitative therapies. These healthy individuals, treated to correct dentofacial deformity, present for surgery with no neurosensory impairment, but yet routinely experience substantial alterations in facial sensation following the surgical procedure. The effects of sensory re-training will be evaluated using three types of outcomes: patient-centered measures to assess the magnitude of the negative effect of altered sensation after surgery and the recovery time needed to reach little or no negative effect; neurosensory behavior measures to assess the patient's ability to learn alternate cues for touch perception and discrimination; and a conventional neurosensory contact threshold measure to assess the actual deficit. Our primary focus will be on the patient's perception of the negative impact of altered sensation on daily life.

ELIGIBILITY:
Inclusion Criteria:

* Developmental dentofacial disharmony
* Receives mandibular advancement by mandibular osteotomy with or without a maxillary procedure.

Exclusion Criteria:

* Congenital anomaly or acute trauma affecting the face.
* Previous facial surgery
* Pregnant at baseline
* Inability to follow written English instructions
* Unwilling to sign informed consent.
* No altered sensation at one week post-surgery
* Altered sensation at baseline reported as numbness or unusual feeling.
* Medical condition associated with systemic neuropathy.

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 186 (Actual)
Dates: Start 2001-12; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Perception of altered sensation
Perception of altered function
Two-point threshold
Two point discrimination
Contact detection

CONTACTS AND LOCATIONS:
Overall Officials: Ceib Phillips, DR, Principal Investigator — Chapel Hill, School of Dentistry
Locations (2):
- United States (2):
  - School of Dentistry, Chapel Hill, North Carolina
  - University Oral and Maxillofacial Surgery, Charlotte, North Carolina